CLINICAL TRIAL: NCT02081027
Title: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Pilot Study of Riluzole for Drug-Refractory Irritability in Autism Spectrum Disorders
Brief Title: Pilot Study of Riluzole for Drug-Refractory Irritability in Autism Spectrum Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CIN001- Riluzole in Autism
Record Dates: First submitted 2013-08-05; First posted 2014-03-07 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Riluzole (Experimental): The maximum dose of riluzole to be used in this study is 200 mg per day divided BID
  Interventions: Drug: Riluzole
- Placebo (Placebo Comparator): Placebo will be administered in the same manner as the riluzole group, in order to maintain subject assignment throughout the study.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Riluzole
  Other Names: Other name: Rilutek
  Arms: Riluzole
Other: placebo
  Arms: Placebo

SUMMARY:
Determine if riluzole shows evidence of efficacy, safety, and tolerability targeting drug-refractory irritability (DRI) in persons with autism spectrum disorders (ASD).

DETAILED DESCRIPTION:
A randomized, double blind, placebo-controlled, 12-week cross-over study (5-week treatment periods with 2-week washout) of adjunctive riluzole in 12 persons with ASD and DRI between the ages of 12 and 25 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 and < 26 years.
* Weight greater than 50 kg.
* Diagnosis of ASD
* Drug-refractory irritability, as defined as screening ABC Irritability subscale (ABC-I) score of ≥18 AND 1) failure of clinically adequate treatment trials of both aripiprazole and risperidone or 2) failure of at least three previous clinically adequate drug trials targeting irritability (one trial must include aripiprazole or risperidone), as confirmed by caregiver reports and medical record review when available.
* Stable dosing of all concomitant psychotropic medications (including those targeting irritability) for four weeks prior to screening visit and during the study.
* Presence of parent/guardian willing to serve as informant for behavioral outcome measures and shipping control sample for Extracellular Signal-Related Kinase biomarker (ERK) assay.

Exclusion Criteria:

* Current use of more than two concomitant psychotropic drugs targeting irritability.
* Current use of valproic acid.
* Current use of drugs with known interaction with riluzole
* Current use of drugs with concomitant glutamatergic or glutamatergic- modulating action medications.
* For female subjects of child bearing potential, a positive serum pregnancy test.
* History of pancreatitis.
* Hemoglobin less than or equal to 8.0 gm/dL.
* Neutropenia with absolute neutrophil count less than or equal to 1.0 K/mcL.
* Problems with kidney functioning, as assessed by lab work
* Any major chronic medical or chronic respiratory illness considered to be uncontrolled by the Principal Investigator.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09-19 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Improvement | Change from baseline to end of week 12
  A clinician-rated global assessment of symptom change rated on a scale from 1 to 7
Aberrant Behavior Checklist- Irritability | Change between baseline and end of each phase
  A parent questionnaire measuring five behavioral domains

CONTACTS AND LOCATIONS:
Overall Officials: Logan Wink, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wink LK, Adams R, Horn PS, Tessier CR, Bantel AP, Hong M, Shaffer RC, Pedapati EV, Erickson CA. A Randomized Placebo-Controlled Cross-Over Pilot Study of Riluzole for Drug-Refractory Irritability in Autism Spectrum Disorder. J Autism Dev Disord. 2018 Sep;48(9):3051-3060. doi: 10.1007/s10803-018-3562-5. PMID 29644582
- See also: Journal of Autism and Developmental Disorders (2018) 48:3051-3060 — https://doi.org/10.1007/s10803-018-3562-5